CLINICAL TRIAL: NCT00490022
Title: The Effect of Dihydrotestosterone (DHT) on Prostate Tissue Androgen Concentrations and Inflammation in Normal Men
Brief Title: Effect of Dihydrotestosterone (DHT) on Prostate Tissue [Short Title: DHT-3]
Acronym: DHT-3
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH); ASCEND Therapeutics (Industry)
Responsible Party: Stephanie T Page, MD, PhD, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31866-A; 1K23AG027238-01A1 (NIH)
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Results first posted 2011-06-09 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Healthy
Keywords: Dihydrotestosterone; Androgen; Prostate
MeSH Terms: interventions — Dihydrotestosterone; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): DHT gel (70 mg/day) for one month
  Interventions: Drug: Dihydrotestosterone (DHT) gel (0.7%)
- 2 (Placebo Comparator): Placebo gel for one month
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Dihydrotestosterone (DHT) gel (0.7%) — DHT gel, 70 mg/day for one month
  Other Names: 17β-Hydroxy-5α-androstane-3-one
  Arms: 1
Drug: Placebo gel — Placebo gel for one month
  Arms: 2

SUMMARY:
The purpose of this research study is to understand the effects of a male hormone normally made in the body called Dihydrotestosterone (DHT) on the prostate gland that is located under the bladder. The knowledge gained from this study may be used to help in the future to develop a safe male hormonal contraceptive to prevent pregnancy, in the safe treatment of low male hormone levels in men, and in the treatment and prevention of diseases of the prostate.

The investigators will be giving DHT in a gel form, to be applied to the skin, or a placebo gel (with no active drug in it). The investigators want to see the effects of DHT on levels of hormones in the blood and in the prostate gland itself. In addition, the investigators will be studying the effects of DHT on the cells and genes expressed within the prostate.

The effect of DHT on the prostate is not known. Some studies suggest blocking production of DHT in the prostate helps growth of the gland with aging (a condition known as benign prostatic hyperplasia, or BPH for short) and may prevent prostate cancer. On the other hand, DHT administration may shrink the prostate, suggesting it may be beneficial for some men. Therefore, further studies looking at the effect of DHT on the prostate are needed.

DETAILED DESCRIPTION:
In this study, we will examine the in vivo effects of DHT supplementation on the prostate and serum inflammatory markers at the molecular level. We hypothesize that increases in serum DHT will not increase intraprostatic DHT or prostate epithelial proliferation, and will be associated with decreases in markers of systemic inflammation. Normal, healthy, male study volunteers will be treated with either placebo gel (Group 1) or DHT gel (Group 2) for one month. Serum hormonal and inflammatory measurements will be assessed before, during, and after treatment, and the relationship between hormones and inflammatory markers associated with cardiovascular risk will be determined. Prostate biopsies will be taken after one month of treatment. Prostate tissue will be analyzed for changes in intraprostatic hormone levels as well as gene expression following treatment.

SPECIFIC AIMS:

1. To determine the effect of increases in serum DHT, without concomitant increases in serum T or estrogen, on intraprostatic androgen levels.
2. To determine the effect of increases in serum DHT, without concomitant increases in serum T or estrogen, on prostate epithelial gene expression.
3. To determine the effect of increases in serum DHT, without concomitant increases in serum T or estrogen, on serum lipids and inflammatory markers including C-Reactive Protein [CRP], Tumor necrosis factor-alpha [TNFα], Interleukin-6 [IL-6], adiponectin, plasminogen activator inhibitor [PAI-I], and leptin.

We will test the hypothesis in normal men (rather than hypogonadal men) as a "proof of principle" investigation. A normal hypothalamic-pituitary-testicular axis and regulation, circulating T and DHT levels and intraprostatic androgen concentrations in healthy, normal men will permit optimal testing of the hypothesis. Exogenous DHT administration in normal men is expected to suppress endogenous gonadotropin and testosterone secretion, compared to more variable effects in hypogonadal men that depend on the degree of hypogonadism in these men and whether they have primary (testicular) or secondary (hypothalamic-pituitary) hypogonadism. Furthermore, intraprostatic T and DHT concentrations and 5 alpha-reductase activity (that is androgen-dependent) is expected to be more variable in hypogonadal men, depending on the degree of androgen deficiency and circulating T and DHT levels. If results in normal men support the hypothesis, subsequent studies could be performed in hypogonadal men. Because of the larger variability in circulating and probably intraprostatic androgen concentrations in hypogonadal men, these studies will require much larger numbers of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males 35-55 years old
* Normal serum total testosterone (300 ng/dl-1000 ng/dl)
* Normal Luteinizing Hormone [LH] and Follicle Stimulating Hormone [FSH] levels
* Informed consent
* Taking no regular medications
* Normal baseline prostate ultrasound, hematology, and liver function tests

Exclusion Criteria:

* History of prostate cancer
* Prostate Specific Antigen [PSA] > 2.0
* American Urological Association [AUA] prostate symptom score > 10
* History of testosterone or anabolic steroid use in the past
* Chronic medical illness or prostate disease
* History of a bleeding disorder or need for anticoagulation
* A first-degree relative (i.e. father, brother) with a history of prostate cancer
* Abnormal digital rectal examination
* Skin condition that might interfere with or be exacerbated by DHT gel use
* History of untreated sleep apnea and/or psychiatric problems
* Participation in another study in the past 2 months
* Participating in a regular physical relationship with a pregnant woman

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2007-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie T Page, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Huggins C, Hodges CV. Studies on prostatic cancer: I. The effect of castration, of estrogen and of androgen injection on serum phosphatases in metastatic carcinoma of the prostate. 1941. J Urol. 2002 Jul;168(1):9-12. doi: 10.1016/s0022-5347(05)64820-3. No abstract available. PMID 12050481
- [Background] Bhasin S, Singh AB, Mac RP, Carter B, Lee MI, Cunningham GR. Managing the risks of prostate disease during testosterone replacement therapy in older men: recommendations for a standardized monitoring plan. J Androl. 2003 May-Jun;24(3):299-311. doi: 10.1002/j.1939-4640.2003.tb02676.x. No abstract available. PMID 12721204
- [Background] Morgentaler A, Bruning CO 3rd, DeWolf WC. Occult prostate cancer in men with low serum testosterone levels. JAMA. 1996 Dec 18;276(23):1904-6. PMID 8968017
- [Background] Schatzl G, Madersbacher S, Thurridl T, Waldmuller J, Kramer G, Haitel A, Marberger M. High-grade prostate cancer is associated with low serum testosterone levels. Prostate. 2001 Apr;47(1):52-8. doi: 10.1002/pros.1046. PMID 11304729
- [Background] Wu FC, von Eckardstein A. Androgens and coronary artery disease. Endocr Rev. 2003 Apr;24(2):183-217. doi: 10.1210/er.2001-0025. PMID 12700179
- [Background] Bagatell CJ, Heiman JR, Matsumoto AM, Rivier JE, Bremner WJ. Metabolic and behavioral effects of high-dose, exogenous testosterone in healthy men. J Clin Endocrinol Metab. 1994 Aug;79(2):561-7. doi: 10.1210/jcem.79.2.8045977.
- [Background] Bartsch W, Klein H, Schiemann U, Bauer HW, Voigt KD. Enzymes of androgen formation and degradation in the human prostate. Ann N Y Acad Sci. 1990;595:53-66. doi: 10.1111/j.1749-6632.1990.tb34282.x. No abstract available. PMID 1695829
- [Background] Bartsch W, Krieg M, Becker H, Mohrmann J, Voigt KD. Endogenous androgen levels in epithelium and stroma of human benign prostatic hyperplasia and normal prostate. Acta Endocrinol (Copenh). 1982 Aug;100(4):634-40. doi: 10.1530/acta.0.1000634. PMID 6181638
- [Background] Page ST, Lin DW, Mostaghel EA, Hess DL, True LD, Amory JK, Nelson PS, Matsumoto AM, Bremner WJ. Persistent intraprostatic androgen concentrations after medical castration in healthy men. J Clin Endocrinol Metab. 2006 Oct;91(10):3850-6. doi: 10.1210/jc.2006-0968. Epub 2006 Aug 1. PMID 16882745
- [Background] Wilson JD. The role of 5alpha-reduction in steroid hormone physiology. Reprod Fertil Dev. 2001;13(7-8):673-8. doi: 10.1071/rd01074. PMID 11999320
- [Background] Andriole GL, Humphrey P, Ray P, Gleave ME, Trachtenberg J, Thomas LN, Lazier CB, Rittmaster RS. Effect of the dual 5alpha-reductase inhibitor dutasteride on markers of tumor regression in prostate cancer. J Urol. 2004 Sep;172(3):915-9. doi: 10.1097/01.ju.0000136430.37245.b9. PMID 15310997
- [Background] Norman RW, Coakes KE, Wright AS, Rittmaster RS. Androgen metabolism in men receiving finasteride before prostatectomy. J Urol. 1993 Nov;150(5 Pt 2):1736-9. doi: 10.1016/s0022-5347(17)35882-2. PMID 7692110
- [Background] Kunelius P, Lukkarinen O, Hannuksela ML, Itkonen O, Tapanainen JS. The effects of transdermal dihydrotestosterone in the aging male: a prospective, randomized, double blind study. J Clin Endocrinol Metab. 2002 Apr;87(4):1467-72. doi: 10.1210/jcem.87.4.8138. PMID 11932266
- [Background] Ly LP, Jimenez M, Zhuang TN, Celermajer DS, Conway AJ, Handelsman DJ. A double-blind, placebo-controlled, randomized clinical trial of transdermal dihydrotestosterone gel on muscular strength, mobility, and quality of life in older men with partial androgen deficiency. J Clin Endocrinol Metab. 2001 Sep;86(9):4078-88. doi: 10.1210/jcem.86.9.7821. PMID 11549629
- [Background] Nelson PS, Clegg N, Arnold H, Ferguson C, Bonham M, White J, Hood L, Lin B. The program of androgen-responsive genes in neoplastic prostate epithelium. Proc Natl Acad Sci U S A. 2002 Sep 3;99(18):11890-5. doi: 10.1073/pnas.182376299. Epub 2002 Aug 16. PMID 12185249
- [Derived] Page ST, Lin DW, Mostaghel EA, Marck BT, Wright JL, Wu J, Amory JK, Nelson PS, Matsumoto AM. Dihydrotestosterone administration does not increase intraprostatic androgen concentrations or alter prostate androgen action in healthy men: a randomized-controlled trial. J Clin Endocrinol Metab. 2011 Feb;96(2):430-7. doi: 10.1210/jc.2010-1865. Epub 2010 Dec 22. PMID 21177791

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 55 normal, healthy men between the ages of 35-55 will be recruited for this study. All subject activities will occur at the University of Washington in Seattle Washington.
Pre-assignment Details: Subjects must meet all study protocol inclusion criteria such as informed consent, normal lab values, normal physical examination and normal prostate ultrasound, and not have exclusion criteria such as a first degree relative with or personal history of prostate cancer, PSA >2.0 or a history of a bleeding disorder or need for anticoagulation.
Groups:
- Placebo DHT Gel: Placebo gel for one month
- DHT Gel: DHT gel (70 mg/day) for one month
Period: Overall Study
Arm/Group | Placebo DHT Gel | DHT Gel
Started | 16 | 15
Completed | 15 | 12
Not Completed | 1 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Subject failed to disclose concommitant | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo DHT Gel | DHT Gel | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44.4 (6.7) | 42.7 (1.6) | 43.6 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 15 | 31
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Prostate Tissue DHT and Testosterone Levels After 28 Days of Treatment With Dihydrotestosterone [DHT] Gel Versus Placebo Gel.
Description: After 4 weeks of either daily dihydrotestosterone transdermal gel or placebo gel, subjects underwent a prostate biopsy. Intraprostatic hormone concentrations, specifically DHT and Testosterone, were measured. Unit of measure is ng/g.
Time Frame: 28-days
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Placebo DHT Gel | DHT Gel
Number analyzed (Participants) | 15 | 12
ng/g
  DHT concentrations | 2.8 (0.2) | 3.1 (0.5)
  Testosterone Concentrations | 0.6 (0.2) | 0.4 (0.1)

2. Secondary Outcome: Prostate Epithelial Cell Proliferation
Description: Prostate epithelial cell proliferation in the prostate biopsy tissue was measured using Ki-67 immunohistochemical staining of prostate epithelium as a marker of cell proliferation (values are number of Ki-67 positive stained cells per 100 prostate epithelial cells). The placebo and treatment groups were compared.
Time Frame: 28-days
Measure: Mean (Standard Deviation); unit: #pos.Ki-67cells per100 prst. epth cells
Arm/Group | Placebo DHT Gel | DHT Gel
Number analyzed (Participants) | 15 | 12
#pos.Ki-67cells per100 prst. epth cells | 1.3 (0.5) | 0.7 (0.9)

ADVERSE EVENTS:
Arm/Group | Placebo DHT Gel | DHT Gel
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/15
Other Adverse Events (participants affected / at risk) | 0/16 | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo DHT Gel (N=16) | DHT Gel (N=15)
Rectal Bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo DHT Gel (N=16) | DHT Gel (N=15)
Urinary Frequency (Renal and urinary disorders) | 0/15 (0) | 1 (1) — Subject experienced urinary frequency. It resolved after discontinuation of DHT gel.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No